CLINICAL TRIAL: NCT07155928
Title: The Effect of Cardiac Rehabilitation on Left Ventricular Remodeling in Patients Undergoing Primary Percutaneous Coronary Intervention for Acute Myocardial Infarction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Muhammad Hatem Hassan Mohammed Maghraby, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR on LV Remod in PPCI Pt
Record Dates: First submitted 2025-08-16; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Acute Myocardial Infarction (AMI); PCI Patients; Percutaneous Coronary Intervention (PCI); Primary Percutaneous Coronary Intervention; Left Ventricle Remodeling
Keywords: Cardiac Rehabilitation; Acute Myocardial Infarction; Primary Percutaneous Coronary Intervention; Left Ventricular Remodeling; Ejection fraction; End-systolic volume; End-systolic diameter; End-diastolic volume; End-diastolic diameter; Functional capacity; Aerobic exercise; Resistance Training
MeSH Terms: conditions — Ventricular Remodeling | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized Control Trial including 2 Parallel Groups
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Standard Treatment + Cardiac Rehabilitation
  Interventions: Behavioral: Cardiac Rehabilitation; Procedure: Primary Percutaneous Coronary Intervention
- Control Group (Active Comparator): Standrad Treatment Only
  Interventions: Procedure: Primary Percutaneous Coronary Intervention

INTERVENTIONS:
Behavioral: Cardiac Rehabilitation — * The cardiac rehabilitation program include supervised exercise training, patient education, and risk factor modification.
  * CR starts 1-3 weeks after PCI (based on the patient's general condition) and lasting 12 weeks thereafter.
  * Patients will undergo a supervised CR program based on published guidelines (FITT principle). The core will be a moderate-intensity aerobic exercise regimen (e.g. treadmill or cycle ergometer) 2-3 times per week for 12 weeks. Each session will last ~20-60 minutes of exercise followed by cool-down, with intensity gradually increased to High intensity interval training (HIIT) in low-moderate risk individuals. Resistance exercises (e.g. light weights or band exercises) will also be included twice weekly. Exercise dose (frequency, intensity, time) will be tracked. Physical therapists will supervise all sessions in an outpatient CR facility or affiliated gym. Patients' vitals and ECG will be monitored during initial sessions for safety.
  Arms: Intervention Group
Procedure: Primary Percutaneous Coronary Intervention — Patients will undergo Primary Percutaneous Coronary Intervention (PPCI) within 24 hours of symptom onset for urgent revascularization of the occluded coronary artery.

SUMMARY:
Cardiac rehabilitation has proven to improve the functional capacity of patients who had acute myocardial infarction. However, its effect on Left ventricular remodeling following an MI event treated with Primary PCI is not yet fully understood. So, for this randomized controlled trial our objectives are as follows:

* Primary: To assess the effect of a structured CR program on LV remodeling parameters (LVEF, LVESV, LVEDV, LVESD, LVEDD + SWMA) in STEMI patients treated with primary PCI.
* Secondary: To evaluate changes in exercise capacity, heart rate recovery and clinical outcomes such as major adverse cardiovascular events and the effect of CR on the patients' Quality of Life.

These results will be compared to the same parameters in a control group that will not undergo cardiac rehabilitation to properly assess the effect of cardiac rehab.

Participants in the intervention group will be asked to undergo a supervised CR program based on published guidelines (FITT principle). The core will be a moderate-intensity aerobic exercise regimen (e.g. treadmill or cycle ergometer) 2-3 times per week for 12 weeks. Each session will last ~20-60 minutes of exercise followed by cool-down, with intensity gradually increased to High intensity interval training (HIIT) in low-moderate risk individuals, as it has shown better improvement in cardiovascular health while being safe in MI patients. Resistance exercises (e.g. light weights or band exercises) will also be included twice weekly. Exercise dose (frequency, intensity, time) will be tracked. Physical therapists will supervise all sessions in an outpatient CR facility or affiliated gym. Patients' vitals and ECG will be monitored during initial sessions for safety.

DETAILED DESCRIPTION:
ST-segment elevation myocardial infarction (STEMI) remains a leading cause of morbidity and mortality worldwide. Primary percutaneous coronary intervention (PCI) is the gold standard for reperfusion therapy in STEMI, significantly improving survival rates. However, adverse left ventricular (LV) remodeling post-STEMI can lead to heart failure, poor clinical outcomes and deterioration in patients' quality of life.

Cardiac rehabilitation (CR) is a multidisciplinary intervention designed to optimize cardiovascular recovery. It involves a spectrum of interventions including a structured exercise program, patient education, nutritional counseling, risk factor modification and psychosocial support. CR is divided into 4 stages. Stage I is in-hospital exercise (early mobilization and patient education). Stage II is early outpatient supervised rehabilitation in rehabilitation centers lasting 3 months post-PCI. Stage III starts at 3-12 months and is usually home-based rehabilitation with frequent visits to rehabilitation centers. Stage IV is long term rehab where the patient continues to exercise and commit to a healthy lifestyle to prevent further episodes of cardiovascular disease. Research has shown that stage II is the most crucial of them all, and starting during early in-hospital setting has shown no further improvement in cardiovascular health.

Exercise-based programs, have especially shown beneficial effects on LV function post-AMI, improving exercise capacity and potentially limiting adverse remodeling process. It has been reported that supervised exercise training after STEMI significantly increased LVEF and reduced the rate of unfavorable remodeling at 6 months compared to usual care.

Moreover, there was a significant reduction in post-treatment LV mass, EF, and LV dimensions relative to pretreatment. It has also been suggested that early initiation of CR may reduce systemic inflammation and promote favorable ventricular remodeling.

However, other studies have shown that CR may not have a clinically significant improvement in LV parameters despite the overall improvement in patient's exercise capacity , but these studies were performed with a small sample size. Other trials have shown mixed results, with some showing favorable remodeling after exercise therapy, and some showing no improvement in cardiac dimensions. Another study mentioned that CR may have a positive effect on LV diastolic dysfunction, without any change to LV dimensions.

As such, the exact impact of CR on LV remodeling specifically in primary PCI-treated STEMI patients requires further clarification, especially with recent evidence highlighting its potential benefits.

Such controversy provides adequate foundation to further research this topic with a larger sample size, inclusion of both sexes, with individualization of exercise protocols based on each patient's tolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Underwent successful primary PCI within 24 hours of symptom onset.
2. Hemodynamically stable and able to participate in rehabilitation.

Exclusion Criteria:

1. Stage IV Heart failure, LVEF < 30%
2. Life-threatening arrhythmias
3. Unstable Angina
4. Severe Valvular Diseases
5. Uncontrolled Hypertension
6. CKD Stages IV and V
7. Hypothyroidism
8. Cardiomyopathy
9. Inability to ambulate or consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in LV remodeling assessed by LV ejection fraction (LVEF) | Before and after a 3-month cardiac rehabilitation program
  LVEF assessed in "%"
Change in LV remodeling assessed by LV end-systolic Volume (LVESV), LV end-diastolic Volume (LVEDV) | Before and after a 3-month cardiac rehabilitation program
  LVESV and LVEDV are both assessed in mL
Change in LV remodeling assessed by LV end-systolic Diameter (LVESD) and LV end-diastolic Diameter (LVEDD). | Before and after a 3-month cardiac rehabilitation program
  LVESD and LVEDD are both assessed in millimeters

SECONDARY OUTCOMES:
Exercise capacity assessed in METs | Before and after a 3-month cardiac rehabilitation program
Heart rate recovery post-exercise. | Before and after a 3-month cardiac rehabilitation program
  HRR is measured in BPM
Incidence of MACE during follow-up | Throughout the 3 month CR program

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy Shams Eddin Mohammad Taher, MD, Study Chair — Assiut University; Magdy Ibrahim Aldesowky Mohamed Algowhary, MD, Study Chair — Assiut University

REFERENCES:
- [Background] Soleimannejad K, Nouzari Y, Ahsani A, Nejatian M, Sayehmiri K. Evaluation of the effect of cardiac rehabilitation on left ventricular diastolic and systolic function and cardiac chamber size in patients undergoing percutaneous coronary intervention. J Tehran Heart Cent. 2014;9(2):54-8. PMID 25861319
- [Background] Scalvini S, Zanelli E, Comini L, Dalla Tomba M, Troise G, Febo O, Giordano A. Home-based versus in-hospital cardiac rehabilitation after cardiac surgery: a nonrandomized controlled study. Phys Ther. 2013 Aug;93(8):1073-83. doi: 10.2522/ptj.20120212. Epub 2013 Apr 18. PMID 23599353
- [Background] Qi Z, Zheng Y, Chan JSK, Tse G, Liu T. Exercise-based cardiac rehabilitation for left ventricular function in patients with heart failure: A systematic review and meta-analysis. Curr Probl Cardiol. 2024 Feb;49(2):102210. doi: 10.1016/j.cpcardiol.2023.102210. Epub 2023 Nov 20. PMID 37993005
- [Background] Mahmoud, S. Y. Z., Mohamed Ahmed; Alamin, Ali Mohamed; Yassin, Ibrahim Abdel-Fattah; and Hassaan, Ahmad Mohammad (2024) (2024). Effect of Cardiac Rehabilitation on Left Ventricular Remodeling After Acute Anterior Wall ST Segment Elevation Myocardial Infarction Treated by Late PCI Using 3D Echocardiography: A Randomized Study. Al-Azhar International Medical Journal, 33. https://doi.org/DOI: https://doi.org/10.58675/2682-339X.2235
- [Background] Dubach P, Myers J, Dziekan G, Goebbels U, Reinhart W, Vogt P, Ratti R, Muller P, Miettunen R, Buser P. Effect of exercise training on myocardial remodeling in patients with reduced left ventricular function after myocardial infarction: application of magnetic resonance imaging. Circulation. 1997 Apr 15;95(8):2060-7. doi: 10.1161/01.cir.95.8.2060. PMID 9133516
- [Background] Ahmed Galal A. Fattah Fahmy MD , Gamal Abdel Hady MD , M. H. H., MD , K. M. M. M. a., & MD, M. E. B. (2021). Continuous Moderate Exercise Influence on Cardiac Remodeling in Patients Underwent Percutaneous Coronary Intervention. SciVision.